CLINICAL TRIAL: NCT00489762
Title: Housing, Heating and Health Study:a Randomised Community Trial
Brief Title: Does Improving Insulation and Heating Improve Health?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Otago (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Heating Study
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Last update posted 2007-06-21 (Estimated); Status verified 2007-06

CONDITIONS: Asthma
Keywords: Childhood; Asthma; Heating; Insulation; Respiratory symptoms
MeSH Terms: conditions — Asthma; Signs and Symptoms, Respiratory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Installation of an energy efficient heater

SUMMARY:
The Housing, Heating and Health Study has enrolled 409 households with ineffective heaters, who have a child with asthma between 6 and 12 years.

In the winter of 2005, houses were insulated and baseline measures taken of indoor temperatures, nitrogen dioxide, with more intensive indoor air quality monitoring in a sub-sample of 33 homes.

Objective data are being collected on the household's health and energy usage. The households randomly assigned to the intervention group will have new heaters installed over the summer.

Results will be available after the follow-up data collection in 2006.

DETAILED DESCRIPTION:
1. Introduction New Zealand houses are relatively poorly constructed and maintained for the temperate climate and most homes are heated to less than the WHO recommended minimum winter temperature of 18°C. Excess winter mortality is comparable to the levels in Portugal and Scotland. The Group's previous Housing, Insulation and Health Study has shown that insulating existing homes leads to a small but significant improvement in health and energy consumption, but raised the question as to whether installing more sustainable heating could increase these gains.
2. Study design

We have enrolled 409 households, who use either plug-in electric heaters or unflued gas heating, and where there is a child with asthma, aged between 6 and 12 years. In the winter of 2005, uninsulated houses were insulated and baseline measures taken of indoor temperatures in the living room and the child's bedroom, and levels of nitrogen dioxide. Intensive monitoring of indoor air quality is being carried out in a sub-sample of 33 homes. All members of the child's family have filled out detailed questionnaires of their health and the heads-of -household have completed a questionnaire on the characteristics of the household's energy usage. Objective measures are also being collected of the household's fuel bills, the child's attendance at school and the family's health care utilisation.

Households are randomised so that the intervention group will have their choice of new, more efficient and sustainable heaters (heat pumps, wood pellet burners, or flued gas heaters) that heat more of the house and which emit no internal emissions installed over the summer. In the winter of 2006, follow-up measures will be taken and then the control households will receive their choice of new heaters.

ELIGIBILITY:
Inclusion Criteria:

* Household has asthmatic child between 6 and 12, is living in study area, and will not be moving in the two years after applying to join the study.

Exclusion Criteria:

* Heating of good quality and comparable to heater that will be installed by the study

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 409 (Actual)
Dates: Start 2005-06; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Asthma Symptoms | One year
FEV1 | One year
Children's days off school and general practitioner visits | One year

SECONDARY OUTCOMES:
Energy usage | One year
Hospitalisation | One year
Temperature in the Home | Four months

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Howden-Chapman, PhD, Study Director — Housing and Health Research Programme
Locations (1):
- University of Otago, Wellington, Wellington Region, New Zealand

REFERENCES:
- [Derived] Gillespie-Bennett J, Pierse N, Wickens K, Crane J, Howden-Chapman P; Housing Heating and Health Study Research Team. The respiratory health effects of nitrogen dioxide in children with asthma. Eur Respir J. 2011 Aug;38(2):303-9. doi: 10.1183/09031936.00115409. Epub 2010 Dec 22. PMID 21177840
- [Derived] Howden-Chapman P, Pierse N, Nicholls S, Gillespie-Bennett J, Viggers H, Cunningham M, Phipps R, Boulic M, Fjallstrom P, Free S, Chapman R, Lloyd B, Wickens K, Shields D, Baker M, Cunningham C, Woodward A, Bullen C, Crane J. Effects of improved home heating on asthma in community dwelling children: randomised controlled trial. BMJ. 2008 Sep 23;337:a1411. doi: 10.1136/bmj.a1411. PMID 18812366
- See also: Click here for more information about the "Housing, Heating and Health Study" on the website of the Housing and Health Research Programme, University of Otago, Wellington — http://www.wnmeds.ac.nz//healthyhousing.html